CLINICAL TRIAL: NCT03829371
Title: A RANDOMIZED, MULTICENTER, OPEN LABEL STUDY COMPARING TWO STANDARD TREATMENTS, BORTEZOMIB-MELPHALAN-PREDNISONE (VMP) WITH OR WITHOUT DARATUMUMAB (Dara-VMP) VS LENALIDOMIDE-DEXAMETHASONE (Rd) WITH OR WITHOUT DARATUMUMAB (Dara-Rd) IN AUTOLOGOUS STEM CELL TRANSPLANTATION (ASCT) INELIGIBLE COMMUNITY POPULATION AFFECTED BY MULTIPLE MYELOMA (MM)
Brief Title: STUDY COMPARING TWO STANDARD TREATMENTS IN AUTOLOGOUS STEM CELL TRANSPLANTATION INELIGIBLE POPULATION AFFECTED BY MULTIPLE MYELOMA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Dr. Alessandra Larocca, Principal Investigator, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Real MM
Record Dates: First submitted 2019-01-22; First posted 2019-02-04 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma
Keywords: TRANSPLANT INELIGIBLE; STANDARD TREATMENTS
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Melphalan; Prednisone; Lenalidomide; Dexamethasone; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ARM A (enrollment closed) (Experimental): Velcade (V):
  * 1.3 mg/m2 subcutaneously on days 1, 4, 8, 11, 22, 25, 29 and 32 in cycles 1-4;
  * 1.3 mg/m2 subcutaneously on days 1, 8, 22 and 29 from cycle 5.
  Melphalan (M):
  - 9 mg/m2 orally on days 1, 2 3 and 4 of each cycle.
  Prednisone (P):
  - 60 mg/m2 orally on days 1, 2, 3 and 4 of each cycle. Each cycle is a 42-day cycle. Duration: Maximum 9 cycles can be performed.
  Interventions: Drug: Velcade; Drug: Melphalan; Drug: Prednisone
- ARM B (enrollment closed) (Experimental): Lenalidomide (R):
  -25 mg orally on days 1-21 of each cycle.
  Dexamethasone (d):
  -40 mg orally on days 1, 8, 15 and 22 of each cycle. Each cycle is a 28-day cycle. Duration: until PD or intolerance.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone
- ARM A2 (Experimental): Velcade (V):
  - 1.3 mg/m2 subcutaneously twice weekly on weeks 1, 2, 4, and 5 of cycle 1 (days 1,4,8,11,22,25,29,32) and once weekly on weeks 1, 2, 4, and 5 of cycles 2 through 9 (days 1,8,22,29).
  Melphalan (M):
  - 9 mg/m2 orally on days 1, 2, 3 and 4 of each cycle.
  Prednisone (P):
  - 60 mg/m2 orally on days 1, 2, 3 and 4 of each cycle.
  Daratumumab:
  -16 mg per kilogram of body weight or 1800 mg Daratumumab subcutaneous (SC) (according to local clinical practice) with oral or intravenous dexamethasone (to manage infusion reactions) at a dose of 20 mg once weekly in cycle 1 (days 1,8,15,22,29,36), every 3 weeks in cycles 2 through 9 (days 1,22), and every 4 weeks thereafter until disease progression or unacceptable toxic effects. Dexamethasone at a dose of 20 mg was substituted for prednisone on day 1 of each cycle.
  Interventions: Drug: Velcade; Drug: Melphalan; Drug: Prednisone; Drug: Daratumumab
- ARM B2 (Experimental): Lenalidomide (R):
  - 25 mg orally on days 1-21 of each cycle.
  Dexamethasone (d):
  - 40 mg orally on days 1, 8, 15 and 22 of each cycle. Each cycle is a 28-day cycles.
  Daratumumab:
  -intravenous at a dose of 16 mg per kilogram of body weight or 1800 mg Daratumumab subcutaneous (SC) (according to local clinical practice) once weekly during cycles 1 and 2, every 2 weeks during cycles 3 through 6, and every 4 weeks thereafter; preinfusion medications were administered approximately 1 hour before each daratumumab dose.
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone; Drug: Daratumumab

INTERVENTIONS:
Drug: Velcade — Subcutaneous use
  Arms: ARM A (enrollment closed); ARM A2
Drug: Melphalan — Oral use
  Arms: ARM A (enrollment closed); ARM A2
Drug: Prednisone — Oral use
  Arms: ARM A (enrollment closed); ARM A2
Drug: Lenalidomide — Oral use
  Arms: ARM B (enrollment closed); ARM B2
Drug: Dexamethasone — Oral use
  Arms: ARM B (enrollment closed); ARM B2
Drug: Daratumumab — Subcutaneous Injection
  Arms: ARM A2; ARM B2

SUMMARY:
Multiple myeloma (MM) is a neoplastic disease deriving from an abnormal proliferation of monoclonal plasma cells in the bone marrow. The survival of MM patients varies from less than 6 months to more than 10 years depending on the stage of disease at diagnosis and prognostic factors. Before 2021, in Italy three current standard treatments were approved for elderly or younger patients with significant comorbidities not eligible for autologous stem cell transplantation (ASCT): bortezomib-melphalan-prednisone (VMP), melphalan-prednisone-thalidomide (MPT) and lenalidomide with low-dose dexamethasone (Rd). Daratumumab is a human IgGk monoclonal antibody that targets CD38, that showed clinical benefit in combination with standard-of-care therapy. The addition of Daratumumab (Dara) to VMP and Rd has created two new standards-of-care regimens Dara-VMP and Dara-Rd, which were approved by the EMA in October 2019, and by the AIFA at the beginning of 2021, based on the results of two large phase 3 studies.

A consistent fraction of elderly patients with cancer and co-morbidities are at increased risk of developing frailty (an emergent geriatric syndrome), as well as physical and cognitive decline, with negative effect on dependance, nutrition and lifestyle, and eventually on responsiveness to and efficacy of treatments.

A frailty scale was recently described that categorized patients with MM as fit, intermediate or frail based on age, comorbidities, and physical and cognitive functioning. The frailty score was a predictor of death, progression of the disease, toxicity and drug discontinuation.

The aim of this study was to compare the first line standard treatments, the triplet VMP versus the doublet Rd, that were available when the study was designed. Until 17th December 2021, 228 patients were enrolled in this trial and randomized to VMP vs Rd. Since Dara-VMP and Dara-Rd have recently become the new standard regimens, in this amendment of the study, daratumumab is added to VMP and Rd.

In this project, we will compare available first line standard treatments, the triplet VMP versus the doublet Rd with or without daratumumab (Dara-VMP, Dara-Rd), in an unselected population of patients ≥ 65 years affected by MM in every day clinical practice.

In the last decade, many novel and expensive drugs have been approved for this disease, yet the general older population is not adequately represented in validating trials. Nevertheless, the results and treatments derived from those registrational trials have often been applied to the real-life older population, with a high risk to produce a negative impact on patient functional capacity and ability to carry out daily tasks, cognitive function, mental status, nutritional condition, social situation/capability to stay at home and finally affecting their quality of life (QoL) and OS.

The main aim of the project is to evaluate the best initial treatment for elderly MM patients and to compare benefits, risks, QoL and costs of currently available, standard treatments according to the patient frailty profile.

DETAILED DESCRIPTION:
All patients will be randomized in a 1:1 ratio to receive:

ARM A (enrollment closed):

Bortezomib (V):

* 1.3 mg/m2 subcutaneously on days 1, 4, 8, 11, 22, 25, 29 and 32 in cycles 1-4;
* 1.3 mg/m2 subcutaneously on days 1, 8, 22 and 29 in cycles 5-9.

Melphalan (M):

- 9 mg/m2 orally on days 1, 2, 3 and 4 of each cycle.

Prednisone (P):

- 60 mg/m2 orally on days 1, 2, 3 and 4 of each cycle. Each cycle is to be repeated every 42 days. Duration: Maximum 9 therapy cycles can be performed. After 9 cycles, patients will be observed until progression disease or the start of a new line of therapy.

ARM A2:

Bortezomib (V) 1. 3 mg/m2 subcutaneously twice weekly on weeks 1, 2, 4, and 5 of cycle 1 (days 1,4,8,11,22,25,29,32) and once weekly on weeks 1, 2, 4, and 5 of cycles 2 through 9 (days 1,8,22,29) Melphalan (M):- 9 mg/m2 orally on days 1, 2, 3 and 4 of each cycle.

Prednisone (P):

- 60 mg/m2 orally on days 1, 2, 3 and 4 of each cycle. Daratumumab (Dara) 16 mg per kilogram of body weight or 1800 mg Daratumumab subcutaneous (SC) (according to local clinical practice) with oral or intravenous dexamethasone (to manage infusion reactions) at a dose of 20 mg once weekly in cycle 1 (days 1,8,15,22,29,36), every 3 weeks in cycles 2 through 9 (days 1,22), and every 4 weeks thereafter until disease progression or unacceptable toxic effects. Dexamethasone at a dose of 20 mg was substituted for prednisone on day 1 of each cycle.

ARM B (enrollment closed):

Lenalidomide (R):

- 25 mg orally on days 1-21 of each cycle.

Dexamethasone (d):

- 40 mg orally on days 1, 8, 15 and 22 of each cycle. Each cycle is a 28-day cycles. Duration: patients will receive treatment until any sign of progression or intolerance.

ARM B2

Lenalidomide (R):

- 25 mg orally on days 1-21 of each cycle.

Dexamethasone (d):

- 40 mg orally on days 1, 8, 15 and 22 of each cycle. Each cycle is a 28-day cycles. Daratumumab (Dara) intravenous at a dose of 16 mg per kilogram of body weight or 1800 mg Daratumumab subcutaneous (SC) (according to local clinical practice) once weekly during cycles 1 and 2, every 2 weeks during cycles 3 through 6, and every 4 weeks thereafter; preinfusion medications were administered approximately 1 hour before each daratumumab dose.

ELIGIBILITY:
Inclusion Criteria:

* Patients has given voluntary written informed consent before the performance of any study related procedure;
* Patients with newly diagnosed symptomatic multiple myeloma (NDMM) based on standard IMWG (International Myeloma Working Group) criteria:
* Clonal bone marrow plasma cells >=10% or biopsy-proven bony or extramedullary plasmacytoma and any one or more of the following CRAB features and myeloma-defining events:
* evidence of end organ damage that can be attributed to the underlying plasma cell proliferative disorder, specifically

  * Hypercalcemia: serum calcium >0.25 mmol/L (>1mg/dL) higher than the upper limit of normal or >2.75 mmol/L (>11mg/dL)
  * Renal insufficiency: creatinine clearance (CLcr)<40 mL per minute (measured or estimated by validated equations) or serum creatinine > 177 micro mol/L (>2mg/dL)
  * Anemia: hemoglobin value of >20g/L below the lower limit of normal, or a hemoglobin value <100g/L
  * Bone lesions: one or more osteolytic lesion on skeletal radiography, CT, or PET/CT. If bone marrow has <10% clonal plasma cells, more than one bone lesion is required to distinguish from solitary plasmacytoma with minimal marrow involvement
* Any one or more of the following biomarkers of malignancy:

  * Clonal bone marrow plasma cell percentage >=60% (clonality should be established by showing kappa/lambda-light-chain restriction on flow cytometry, immunohistochemistry, or immunofluorescence. Bone marrow plasma cell percentage should preferably be estimated from a core biopsy specimen; in case of a disparity between the aspirate and core biopsy, the highest value should be used)
  * Involved:uninvolved serum free light chain ratio >=100 (values based on the serum Freelite assay. The involved free light chain must be >=100 mg/L)
  * >1 focal lesion detected by MRI (magnetic resonance imaging) studies (each focal lesion must be 5 mm or more in size
* According to physician's opinion, patients can undergo either one of the two standard treatments and procedures;
* Females of childbearing potential (FBCP) must use an effective contraceptive method for 28 days before the study treatment, during the treatment and for at least 3 months after the last dose of study drugs;
* Male subjects must use an effective barrier method if sexually active with FCBP during treatment and for at least 6 months after the last dose of study drug;
* Patients should be ineligible for ASCT, defined as:
* >= 65 years old
* younger than 65 years but who reject the transplant procedure or with abnormal cardiac, pulmonary, hepatic and renal function defined as [1]:

  * LVEF (left ventricular ejection fraction) < 40%
  * FEV1 (forced expiratory volume-1 second) < 40%
  * Bilirubin > 1.5 UNL, AST/ALT >2.5 UNL Creatinine clearance < 60 mL/min.

Exclusion Criteria:

* Hypersensitivity to any active substance or to any of the excipients (lactose, microcrystalline cellulose, croscarmellose sodium, magnesium stearate, boron, mannitol, nitrogen, crospovidone, colloidal anhydrous silica, hypromellose, titanium dioxide, macrogol, talc, sodium starch glycolate, sodium benzoate, propylene glycol, sodium dihydrogen phosphate, hydroxypropyl beta cyclodextrin, sodium saccharin, sodium EDTA, sodium hydroxide, L-histidine, L-histidine hydrochloride monohydrate, L-methionine, polysorbate 20, sorbitol (E420), recombinant human hyaluronidase (rHuPH20));
* Hereditary intolerance to fructose;
* Pregnant and lactating women;
* FBCP that do not follow the Pregnancy Prevention Plan requirements;
* Acute diffuse infiltrative pulmonary and pericardial disease;
* Acute viral infections (e.g. herpes simplex or ocular herpes simplex, herpes zoster, varicella);
* Systemic mycotic or bacterial infections, unless specific anti-infectious therapy is ongoing;
* Peptic ulcer;
* Psychosis;
* Administration of prophylactic vaccine from 8 to 2 weeks before starting treatment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2027-01-03 (Estimated); Study Completion 2030-01-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 5 years
  Number of months from the date of randomization to the date of first observation of PD, or death from any cause as an event.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 5 years
  Overall response rate will include complete response (CR), very good partial response (VGPR) and partial response (PR) using the International Response Criteria. Responders are defined as subjects with at least a PR.
Duration of response (DOR) | 5 years
  Time between first documentation of response and PD. Responders without disease progression will be censored either at the time of lost to FU, at the time of death due to other cause than PD, or at the end of the study.
Overall survival (OS) | 5 years
  Time between randomization and death. Subjects who die will be censored at time of death as an event, regardless cause of death.
Progression-free survival 2 (PFS2) | 5 years
  Time from randomization to objective tumor progression on next-line treatment or death from any cause.
Time to next therapy (TNT) | 5 years
  Time to next therapy will be measured from the date of randomization to the date of next anti-myeloma therapy. Death due to any cause before starting therapy will be considered an event.
Time to progression (TTP) | 5 years
  Time to progression will be measured from the date of randomization to the date of first observation of PD, or deaths related to PD.
Adverse events | 5 years
  Safety will be evaluated by assessing the incidence, severity and type of AEs according to NCI-CTCAE v. 4.0.
Rate of treatment discontinuation or death for toxicity | 5 years
  Incidence of treatment discontinuation for toxicities as well as the rate of death for toxicity will be evaluated during the entire duration of the trial (toxicities evaluated according to NCI-CTCAE v. 4.0)
Frailty score | 5 years
  Validation of Myeloma Frailty Score (fit score=0; intermediate-fitness score=1, and frail score≥2) that assess comorbidities, cognitive and physical status in real population according to geriatric assessment and considering patients' non-Myeloma polydrug therapies.
Quality of Life through Health-Related QoL (HRQoL) | 5 years
  Quality of Life will be evaluated through questionnaire: EORTC-QLQ-C30 (a generic, multidimensional, cancer-specific QoL questionnaire).
Quality of Life through Health-Related QoL (HRQoL) | 5 years
  Quality of Life will be evaluated through questionnaire for MM patients: QLQ-MY20 (a specific 20- item MM module).
Quality of Life through Health-Related QoL (HRQoL) | 5 years
  Quality of Life will be evaluated through questionnaire: EQ-5D-5L (a generic assessment of five health categories and overall health score).
Direct health related costs and indirect costs | 5 years
  Health-related costs will be reported through Questionnaires For Patients Costs Evaluation reported in the protocol evaluating working activities.
Direct health related costs and indirect costs | 5 years
  Health-related costs will be reported through Questionnaires For Patients Costs Evaluation reported in the protocol evaluating care assistance.
Direct health related costs and indirect costs | 5 years
  Health-related costs will be reported through Questionnaires For Patients Costs Evaluation reported in the protocol evaluating health care visit.
Risk of infectious complications | 5 years
  Infectious risk complications will be evaluated through a scale evaluating the number of adverse events, severity, type of infection, need for hospitalization (yes/no), number of days of suspension of study treatment. All these data will be combined in the statistical analysis to combine different outcome of treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento di Biotecnologie Molecolari e Scienze per la Salute, Torino, TO, Italy

IPD SHARING:
Plan to Share IPD: Undecided